CLINICAL TRIAL: NCT04054050
Title: Bright Light Therapy for Sleep Disturbance in People With Multiple Sclerosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00222887; R03HD101056 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: sleep disturbance; insomnia; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Parasomnias; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Light therapy (Experimental): Participants receive one hour of morning (within 9:00am-11:00am) and afternoon/evening (within 5:00pm-7:00pm).
  Interventions: Other: Light therapy

INTERVENTIONS:
Other: Light therapy — Bright light (10,000 lux) therapy will be administered via a light box.

SUMMARY:
Sleep disturbance is common in people with multiple sclerosis (MS) and contributes to diminished quality of life. Bright light therapy may be an innovative strategy to reduce sleep disturbance in MS, possibly through its effects on a subtype of retinal ganglion cells that help regulate circadian rhythms and sleep. This pilot study will evaluate whether, in people with MS, bright light therapy reduces sleep disturbance and explore whether light therapy improves function of these cells.

DETAILED DESCRIPTION:
Multiple sclerosis (MS), an inflammatory and neurodegenerative disorder of the central nervous system (CNS), is the most common cause of progressive neurologic dysfunction in early to middle adulthood. People with MS are a markedly high risk for sleep disturbance. Estimates of the lifetime prevalence of sleep disturbance in MS reach 50%; sleep disturbance is also associated with excess MS-associated morbidity and diminished quality of life. Despite the high burden of impaired sleep and its contribution to adverse MS outcomes, effective approaches to treat and ameliorate disturbed sleep in people with MS remain poorly understood. There is unmet need to develop safe and effective rehabilitative alternatives to mitigate sleep disturbance in MS. Prior research supports the use of timed bright light therapy (LT) as one such approach for insomnia and sleepiness in those with sleep disorders or other neurologic diseases. Yet, the safety and potential effectiveness of timed LT have yet to be tested in MS. The goal of the proposed study is to conduct a detailed intervention study testing if timed bright LT in people with MS is 1) safe (primary outcome) and 2) potentially effective for reducing sleep disturbance (specifically, reducing insomnia, fatigue and improving sleep efficiency, quantity and quality as secondary outcomes). The study will also explore whether LT stimulates a novel subtype of retinal ganglion cells which are central to the regulation of circadian rhythms and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* Evidence of sleep disturbance
* Stable on immunomodulatory MS therapy or no therapy for at least 6 months prior to study initiation
* Stable on antidepressants for at least 3 months prior to study initiation and no evidence
* Stable on fatigue medication for at least 3 months prior to study initiation
* Willing and able to provide informed consent and follow study procedures.

Exclusion Criteria:

* Evidence of cognitive impairment
* Low risk for sleep disordered breathing
* Other comorbid ophthalmologic disorders (e.g. cataracts, glaucoma, blindness)
* Traveled across two time zones within 90 days of study screening.
* Not participating in shift work
* MS relapse or history of acute optic neuritis within 30 days
* No prior history of bipolar disorder
* No evidence of current depression
* Diagnosis of severe periodic limb movement disorder or severe restless legs syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 2 weeks
  The number of adverse events will be documented and categorized by organ system

SECONDARY OUTCOMES:
Change in sleep quantity as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 weeks
  The PSQI has a sub-component that quantifies sleep quantity. The investigators will assess change in sleep quantity (difference in minutes) as assessed by this sub-component.
Change in sleep efficiency as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 weeks
  The PSQI has a sub-component that quantifies sleep efficiency. The investigators will assess change in sleep efficiency (difference in minutes) as assessed by this sub-component.
Change in overall sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 weeks
  The PSQI has an overall score that ranges from 0 to 21. The investigators will assess change in the overall PSQI score.
Change in sleep efficiency as assessed by actigraphy | Baseline, 2 weeks
  Change in sleep efficiency is calculated as time sleeping divided by time in bed which is measured by actigraphy.
Change in total sleep time | Baseline, 2 weeks
  Change in total sleep time (minutes) as quantified by actigraphy
Change in insomnia severity as assessed by the Insomnia Severity Index (ISI) | Baseline, 2 weeks
  The ISI is validated questionnaire assessing insomnia from which a total score is calculated and ranges from 0 to 28. The investigators will calculate change in the overall ISI score.
Change in daytime sleepiness as assessed by the Epworth Sleepiness Scale (ESS) | Baseline, 2 weeks
  The ESS is validated questionnaire assessing daytime sleepiness from which a total score is calculated and ranges from 0 to 24. The investigators will calculate change in the overall ESS score.
Change in fatigue severity as assessed by the Neuro-QoL fatigue questionnaire | Baseline, 2 weeks
  The Neuro-QoL fatigue severity score (short form) is a validated 8-question assessment of fatigue from which T-scores ranging from 0 to 100 can be obtained. The investigators will assess change in Neuro-QoL fatigue severity.
Change in function of intrinsically photosensitive retinal ganglion cells | Baseline, 2 weeks
  Change in function of intrinsically photosensitive retinal ganglion cells as quantified by the relative change in pupillary light response to blue light.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn C Fitzgerald, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers. Since the study will enroll only 24 individuals, even if stripped of identifiers, it may still be possible to identify participants. Thus, data will not be shared.